CLINICAL TRIAL: NCT00963911
Title: Validation of a Screening Tool in Geriatric Oncology
Acronym: ONCODAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IB 2008-06; IB-ONCODAGE (Other: Insitut Bergonie); IB 2008-06 (Other: Insitut Bergonie); 2008-A00322-53 (Other: AFSSAPS)
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer; Colorectal Cancer; Head and Neck Cancer; Lung Cancer; Lymphoma; Prostate Cancer
Keywords: colon cancer; rectal cancer; non-small cell lung cancer; small cell lung cancer; hypopharyngeal squamous cell carcinoma; laryngeal squamous cell carcinoma; laryngeal verrucous carcinoma; lip and oral cavity squamous cell carcinoma; oral cavity verrucous carcinoma; nasopharyngeal squamous cell carcinoma; oropharyngeal squamous cell carcinoma; paranasal sinus and nasal cavity squamous cell carcinoma; salivary gland squamous cell carcinoma; prostate cancer; breast cancer; adult non-Hodgkin lymphoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Lymphoma; Prostatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Squamous Cell Carcinoma of Head and Neck; Lymphoid Interstitial Pneumonia; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Included patients (Experimental): Screening tests (G8 and VES-13)
  Interventions: Other: Geriatric screening tests; Other: Multidimensional geriatric assessment

INTERVENTIONS:
Other: Geriatric screening tests — The G-8 consists of eight items: patient age (>85, 80-85, <80), and seven items from the original 18-item MNA (Mini Nutritional Assessment: appetite changes, weight loss, mobility, neuropsychological problems, body mass index, medication, and self-rated health). The total score ranges from 0 to 17, with lower scores indicating a higher risk of impairments. The cut-off value for an 'impaired' reference test score was <=14 and the time taken to complete the test was recorded.
  VES-13 is a self-administered questionnaire that was completed during the first visit after enrollment. For three pre-identified centers, patients also filled in the questionnaire at the following geriatric visit. VES-13 consisted of four groups of questions: age, self-perceived health, difficulties to perform six specific activities, and difficulties to perform daily living tasks due to health concerns. The score ranged from 0 to 10 and a score >=3 was considered to show impairment.
  Other Names: G-8
Other: Multidimensional geriatric assessment — Patients underwent a geriatric evaluation in the month following the completion of G8 and VES-13 (+/- seven days) before treatment began. The nurse completed six of the seven instruments of the MGA (MNA, Timed Get up and Go (TUG), Activities of Daily Living (ADL), Instrumental ADL (IADL), Mini Mental State Examination (MMSE), and Geriatric Depression Scale (GDS-15)), and the geriatrician rated comorbidity on the Cumulative Illness Rating Scale (CIRS-G), recorded the time required for the consultation, identified patients who needed personalized geriatric interventions, and, if necessary, proposed further geriatric evaluation (outside of the scope of this study).
  Other Names: MGA

SUMMARY:
RATIONALE: A screening questionnaire may help doctors plan better treatment for older patients with cancer.

PURPOSE: This clinical trial is studying a questionnaire in screening older patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Validate a new screening tool (G8).

Secondary

* Validate the French version of the screening tool "Vulnerable Elders Survey (VES-13)".
* Evaluate the merits of the screening tools (G8 and VES-13).
* Assess the screening tool in specific populations.
* Assess the number and type of interventions proposed after thorough geriatric assessment.
* Compare the two new tools (G8 vs VES-13).

OUTLINE: This is a multicenter study.

During the first consultation, patients have an initial clinical evaluation questionnaire comprising the G8. They also complete the self-questionnaire VES-13. Within 30 days, patients have a thorough geriatric assessment, including quality of life and physical function, by a physician without access to the G8 or VES-13 questionnaires. A blood specimen is also collected.

Information on health status and quality of life is collected from medical records or from the doctor after 1 and 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cancer including the following types:

  * Colon
  * Rectal
  * Lung
  * Squamous cell carcinoma of the head and neck
  * Breast
  * Prostate
  * Non-Hodgkin lymphoma
* Planning to undergo first-time treatment comprising medicine, surgery, or radiotherapy

PATIENT CHARACTERISTICS:

* No persons deprived of liberty or under guardianship
* No psychological, familial, social, or geographical reasons that would make monitoring clinically impossible

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1674 (Actual)
Dates: Start 2008-08-05 (Actual); Primary Completion 2010-03-08 (Actual); Study Completion 2015-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Soubeyran, MD, PhD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellera CA, Artaud F, Rainfray M, Soubeyran PL, Mathoulin-Pelissier S. Modeling individual and relative accuracy of screening tools in geriatric oncology. Ann Oncol. 2017 May 1;28(5):1152-1157. doi: 10.1093/annonc/mdx068. PMID 28327973
- [Result] Soubeyran P, Bellera C, Goyard J, Heitz D, Cure H, Rousselot H, Albrand G, Servent V, Jean OS, van Praagh I, Kurtz JE, Perin S, Verhaeghe JL, Terret C, Desauw C, Girre V, Mertens C, Mathoulin-Pelissier S, Rainfray M. Screening for vulnerability in older cancer patients: the ONCODAGE Prospective Multicenter Cohort Study. PLoS One. 2014 Dec 11;9(12):e115060. doi: 10.1371/journal.pone.0115060. eCollection 2014. PMID 25503576

RESULTS

PARTICIPANT FLOW:
Groups:
- Included Patients: Patients older than 70 years
Period: Overall Study
Arm/Group | Included Patients
Started | 1674
Completed | 1674
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is restricted to eligible patients only.
Groups:
- Eligible Patients: Patients older than 70 years and were included either before any first-line treatment, or between any two steps of a pre-defined first-line treatment sequence (chemotherapy, endocrine therapy, targeted treatment, surgery or radiotherapy) for various types of histologically-confirmed cancer (colon, lung, upper aero digestive tract (UAT)/head and neck, breast, prostate, and non-Hodgkin's lymphomas (NHL)).
Arm/Group | Eligible Patients
Number analyzed (Participants) | 1597
Age, Customized [Count of Participants; unit: Participants]
  70-74 years | 493
  75-79 years | 481
  80-84 years | 392
  85 years and older | 231
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1110
  Male | 487
Region of Enrollment [Number; unit: participants]
  France | 1597

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of the G8 Questionnaire
Description: Sensitivity of the G8 questionnaire measured as Percentage of Participants with a Positive G8 among patients with a positive MGA. The G8 consists of eight items: patient age (>85, 80-85, <80), and seven items from the original 18-item MNA (Mini Nutritional Assessment: appetite changes, weight loss, mobility, neuropsychological problems, body mass index, medication, and self-rated health). The total score ranges from 0 to 17, with lower scores indicating a higher risk of impairments. The cut-off value for an 'impaired' reference test score was <=14.
  Multidimensional geriatric assessment (MGA): Patients underwent a geriatric evaluation in the month following the completion of VES-13. The nurse completed six instruments of the MGA (MNA, Timed Get up and Go, Activities of Daily Living (ADL), Instrumental ADL, Mini Mental State Examination, and Geriatric Depression Scale, and the geriatrician rated comorbidity on the Cumulative Illnes Rating Scale.
Time Frame: at inclusion (at completion of the G8 questionnaire)
Population: Eligible patients assessable for the primary outcome measure AND with a positive MGA
Measure: Number (95% Confidence Interval); unit: % of Participants with a positive G8
Groups:
- Eligible Patients Assessable for the Primary Outcome Measure: Patients older than 70 years and included either before any first-line treatment, or between any two steps of a pre-defined first-line treatment sequence (chemotherapy, endocrine therapy, targeted treatment, surgery or radiotherapy) for various types of histologically-confirmed cancer (colon, lung, upper aero digestive tract (UAT)/head and neck, breast, prostate, and non-Hodgkin's lymphomas (NHL)), and for whom G8 as well as at least one instrument of the multidimensional assessment were available.
Arm/Group | Eligible Patients Assessable for the Primary Outcome Measure
Number analyzed (Participants) | 1151
% of Participants with a positive G8 | 76.5 [73.9 to 78.9]

2. Secondary Outcome: Specificity of the G8 Questionnaire
Description: Specificity of the G8 questionnaire measured as percentage of participants with a negative G8 test among patients with a negative MGA.The G8 consists of eight items: patient age (>85, 80-85, <80), and seven items from the original 18-item MNA (Mini Nutritional Assessment: appetite changes, weight loss, mobility, neuropsychological problems, body mass index, medication, and self-rated health). The total score ranges from 0 to 17, with lower scores indicating a higher risk of impairments. The cut-off value for an 'impaired' reference test score was <=14.
  Multidimensional geriatric assessment (MGA): Patients underwent a geriatric evaluation in the month following the completion of VES-13. The nurse completed six instruments of the MGA (MNA, Timed Get up and Go, Activities of Daily Living (ADL), Instrumental ADL, Mini Mental State Examination, and Geriatric Depression Scale, and the geriatrician rated comorbidity on the Cumulative Illnes Rating Scale.
Time Frame: at inclusion (at completion of the G8 questionnaire)
Population: Eligible patients assessable for the primary outcome measure AND with a negative MGA
Measure: Number (95% Confidence Interval); unit: % of Participants with a negative G8
Arm/Group | Eligible Patients Assessable for the Primary Outcome Measure
Number analyzed (Participants) | 284
% of Participants with a negative G8 | 64.4 [58.6 to 70.0]

3. Secondary Outcome: Sensitivity of the VES-13 Questionnaire
Description: Sensitivity of the VES-13 questionnaire measured as percentage of participants with a positive VES-13 test among patients with a positive MGA. VES-13 is a self-administered questionnaire that was completed during the first visit after enrollment. For 3 pre-identified centers, patients filled in the questionnaire at the following geriatric visit. VES-13 consisted of 4 groups of questions: age, self-perceived health, difficulties to perform 6 specific activities, and difficulties to perform daily living tasks due to health concerns. The score ranged from 0 to 10 and a score >=3 was considered to show impairment.
  Multidimensional geriatric assessment (MGA): see measure description for primary outcome.
Time Frame: at inclusion
Population: Eligible Patients Assessable for the Primary Outcome Measure AND with a positive VES-13
Measure: Number (95% Confidence Interval); unit: % of Participants with a positive VES13
Arm/Group | Eligible Patients Assessable for the Primary Outcome Measure
Number analyzed (Participants) | 1151
% of Participants with a positive VES13 | 68.7 [66.0 to 71.4]

4. Secondary Outcome: Specificity of the VES-13 Questionnaire
Description: Specificity of the VES-13 questionnaire measure as the percentage of participants with a negative VES-13 test among patients with a negative MGA. VES-13 is a self-administered questionnaire that was completed during the first visit after enrollment. For 3 pre-identified centers, patients filled in the questionnaire at the following geriatric visit. VES-13 consisted of 4 groups of questions: age, self-perceived health, difficulties to perform 6 specific activities, and difficulties to perform daily living tasks due to health concerns. The score ranged from 0 to 10 and a score >=3 was considered to show impairment.
  Multidimensional geriatric assessment (MGA): see measure description for primary outcome.
Time Frame: at inclusion (at completion of the G8 questionnaire)
Population: Eligible patients assessable for the primary endpoint (sensitivity of the G8 questionnaire) and with a negative MGA
Measure: Number (95% Confidence Interval); unit: % of Participants with a negative VES13
Arm/Group | Eligible Patients Assessable for the Primary Outcome Measure
Number analyzed (Participants) | 284
% of Participants with a negative VES13 | 74.3 [68.8 to 79.3]

5. Secondary Outcome: Reproducibility of the G8 Questionnaire
Description: Reproducibility of G8 was assessed by comparing the score on the actual G8 with the scores extracted from the corresponding seven questions of MNA completed during the MGA for all patients. The G8 consists of eight items: patient age (>85, 80-85, <80), and seven items from the original 18-item MNA (Mini Nutritional Assessment: appetite changes, weight loss, mobility, neuropsychological problems, body mass index, medication, and self-rated health). The total score ranges from 0 to 17, with lower scores indicating a higher risk of impairments. The cut-off value for an 'impaired' reference test score was <=14.
Time Frame: at inclusion (at completion of the G8 questionnaire)
Population: Eligible Patients Assessable for the Primary Outcome Measure AND with two assessments of the G8 available
Measure: Number (95% Confidence Interval); unit: Kappa coefficient of correlation
Arm/Group | Eligible Patients Assessable for the Primary Outcome Measure
Number analyzed (Participants) | 1429
Kappa coefficient of correlation | 0.65 [0.61 to 0.70]

6. Secondary Outcome: Reproducibility of the VES-13 Questionnaire
Description: Reproducibility of VES-13 was assessed based on a subgroup of patients included in three pre-identified centers who completed the questionnaire on two occasions. VES-13 is a self-administered questionnaire that was completed during the first visit after enrollment. For 3 pre-identified centers, patients filled in the questionnaire at the following geriatric visit. VES-13 consisted of 4 groups of questions: age, self-perceived health, difficulties to perform 6 specific activities, and difficulties to perform daily living tasks due to health concerns. The score ranged from 0 to 10 and a score >=3 was considered to show impairment.
Time Frame: at inclusion (at completion of the G8 questionnaire)
Population: Eligible Patients Assessable for the Primary Outcome Measure AND with two assessments of the VES-13 available
Measure: Number (95% Confidence Interval); unit: Kappa coefficient of correlation
Arm/Group | Eligible Patients Assessable for the Primary Outcome Measure
Number analyzed (Participants) | 251
Kappa coefficient of correlation | 0.64 [0.54 to 0.73]

ADVERSE EVENTS:
Time Frame: at baseline (at completion of the G8 questionnaire)
Groups:
- Included Patients: Screening tests (G8 and VES-13)
  The G-8 consists of eight items: patient age (>85, 80-85, <80), and seven items from the original 18-item MNA (Mini Nutritional Assessment: appetite changes, weight loss, mobility, neuropsychological problems, body mass index, medication, and selfrated health). The total score ranges from 0 to 17, with lower scores indicating a higher risk of impairments. The cut-off value for an 'impaired' reference test score was <=14.
  VES-13 is a self-administered questionnaire that was completed during the first visit after enrollment. For three pre-identified centers, patients also filled in the questionnaire at the following geriatric visit. VES-13 consisted of four groups of questions: age, self-perceived health, difficulties to perform six specific activities, and difficulties to perform daily living tasks due to health concerns. The score ranged from 0 to 10 and a score >=3 was considered to show impairment.
  Multidimensional geriatric assessment: Patients underwent a geriatric evaluation in the month following the completion of G8 and VES-13 (+/- seven days) before treatment began. The nurse completed six of the seven instruments of the MGA (MNA, Timed Get up and Go (TUG), Activities of Daily Living (ADL), Instrumental ADL (IADL), Mini Mental State Examination (MMSE), and Geriatric Depression Scale (GDS-15)), and the geriatrician rated comorbidity on the Cumulative Illness Rating Scale (CIRS-G).
Arm/Group | Included Patients
All-Cause Mortality (participants affected / at risk) | 0/1674
Serious Adverse Events (participants affected / at risk) | 0/1674
Other Adverse Events (participants affected / at risk) | 0/1674

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes